CLINICAL TRIAL: NCT06011564
Title: eDENT Oral Health- the Gateway to Quality of Care and Everyday Life at Old Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Blekinge Institute of Technology (Other)
Collaborators: Kristianstad University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BTH-6.1.1-0059-2016
Record Dates: First submitted 2023-06-12; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Mild Cognitive Impairment; Gingivitis; Periodontal Diseases
Keywords: Mild Cognitive Impairment; Oral Health; Quality of Life
MeSH Terms: conditions — Cognitive Dysfunction; Gingivitis; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Reminder function
  Interventions: Device: Reminder function on Android computer tablet
- control (No Intervention): No reminder

INTERVENTIONS:
Device: Reminder function on Android computer tablet — Computer tablet with reminder function
  Arms: Intervention

SUMMARY:
The investigators will present a new strategy for working with oral health for the group of elderly people with various degrees of mild cognitive impairments. The investigators hope that by introducing a powered toothbrush with functions that make it possible to remind and gather information about the use, the investigators will primarily facilitate oral care for this group, and are proposing that this will lead to higher quality of life of the persons involved.

DETAILED DESCRIPTION:
The investigators will present a new strategy for working with oral health for the group of elderly people with various degrees of mild cognitive impairments. The investigators hope that by introducing a powered toothbrush with functions that make it possible to remind and gather information about use, the investigators will primarily facilitate oral care for this group, and are proposing that this will lead to higher quality of life of the persons involved. Secondarily this will have great impact on the care/carer situation as well as the need for reactive dental care. Expected results is to see both how the actual reminders can be designed in order to accommodate for this group, the context of how these reminders can be used and ultimately if this has an impact on oral health for the group of elderly people with various degrees of mild cognitive impairments.

With age, functional decline occurs and the incidence and prevalence of chronic diseases increase, so aging is an important risk for developing medical conditions. Along with age, the prevalence of dementia increases significantly.

Persons with dementia show a higher prevalence of coronal and root caries and present more often with root remnants as the utilization of dental services becomes scarce. Patients with dementia had an increased likelihood of tooth loss and untreated caries, as well as

presenting with poor oral and denture hygiene compared with non-demented persons. In the initial stages of the disease, this condition may be related to a shift in priorities and a reluctance to brush the teeth. In addition, there is the inability to accurately perform oral hygiene measures due to poor motor skills and sacropenia, especially of the hand-grip strength, render oral hygiene measures more difficult to perform. When the disease progresses, patients will become increasingly dependent on supervision/assistance on oral hygiene procedures. Co-operation is required when a carer has to perform oral hygiene measures and access to the mouth has to be granted. Poor oral hygiene and the presence of abundant biofilm fosters periodontal disease and caries. Combined with a shift in dietary intake towards more sweet food-stuffs the risk factors for developing carious lesions increases significantly. The risk of caries is further increased as result of a decreased salivary flow due to medication intake.

Previous research has demonstrated that the use of a powered toothbrush instead of a manual one reduces plaque and gingivitis more effectively than manual toothbrushes . The reduction of gingivitis using an electric toothbrush as compared to a manual one is reported to be in the range of 11 to 17%. According to the American Dental association tooth brushing should be performed twice daily for two minutes each time. On average it is estimated that people brush their teeth for less than a minute per day. The efficacy of a toothbrush is highly dependent on how long time the individual is actually using the device and it can be anticipated that individuals with mild cognitive impairment may forget to use the tooth brush on a daily basis and also that whenever using the brush the time spent may be even shorter than 30 seconds each time. The control group will be supplied with a powered toothbrush only and instructed to use any other means of tooth cleaning (ie. interdental cleaning) as before. It is anticipated that a temporary improvement of oral hygiene will occur in the control group, but the temporary improvement may not be sustainable among individuals with mild cognitive impairment. Accordingly, there will not be an added benefit for either the individual or the society only to supply individuals with cognitive impairment with a powered toothbrush.

In the test group, individuals are supplied with a powered toothbrush and a tablet with reminder functions. It is anticipated that the brush will be used more frequently and possibly also for longer periods compared to the group without such reminder functions, resulting in >30% improvement compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Being 55 years or older
* Having experienced memory problems in the last six months before inclusion
* Having a Mini-Mental State Examination score of 20-28
* Are not receiving any formal care
* Having at least ten teeth of their own

Exclusion Criteria:

* Having a terminal illness with less than three years of expected survival
* Having another known significant cause of disease explaining cognitive impairment

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Change in the amount of dental plaque | From baseline, to month 6, and to month 12, and to month 24, and to month 36
  Presence of dental plaque measured on four of the tooth surfaces presented as a percentage
Change in the amount of gingival bleeding on probing | From baseline, to month 6, and to month 12, and to month 24, and to month 36
  Number of bleeding from the gingiva measured on four sides of the teeth presented as a percentage
Change in the number of periodontal pockets 4 mm or deeper | From baseline, to month 6, and to month 12, and to month 24, and to month 36
  The number of periodontal pockets 4 mm or deeper measured on four of the tooth surfaces presented as a percentage
Change in values for the quality of life instrument QoL-AD | From baseline, to month 6, and to month 12, and to month 24, and to month 36
  The value for the quality of life instrument QoL-AD (Quality of Life Alzheimer Disease) is measured on a scale from 0-30, where 30 corresponds to the highest quality of life
Change in values for the oral health related quality of life instrument OHIP-14 | From baseline, to month 6, and to month 12, and to month 24, and to month 36
  The value for the oral health-related quality of life instrument OHIP-14 (Oral Health Impact Profile-14) is measured on a scale from 0-56 where 0 corresponds to the highest quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Johan Sanmartin-Berglund, Professor, Study Chair — Blekinge Institute of Technology
Locations (1):
- Blekinge Institute of Technology, Karlskrona, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The trial protocol and the datasets used and analyzed during the current study are available upon reasonable request.
Supporting Information: Study Protocol
Time Frame: From 2023-06-12
Access Criteria: The trial protocol and the datasets used and analyzed during the current study are available upon reasonable request.